CLINICAL TRIAL: NCT00812097
Title: Study of the Safety and Effectiveness of Mentor Siltex® Contour Profile Gel Mammary Prostheses in Patients Who Are Undergoing Primary Breast Augmentation,Primary Breast Reconstruction or Revision
Brief Title: Mentor Siltex® Contour Profile Gel Mammary Prosthesis Clinical Trial
Acronym: CPG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A105-0601-4
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Revision
Keywords: Breast Augmentation; Breast Reconstruction; Breast Revision; Silicone gel; Contour Profile Gel; Siltex®

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Primary Augmentation (Other): The Primary Augmentation cohort will include patients who wish general breast enlargement receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants.
  Interventions: Device: Mentor Siltex® Contour Profile Gel Mammary Prosthesis
- Primary Reconstruction (Other): The Primary Reconstruction cohort will include patients with loss of breast due to mastectomy or with deformities secondary to disease, malignancy, trauma, and congenital deformity receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants.
  Interventions: Device: Mentor Siltex® Contour Profile Gel Mammary Prosthesis
- Revision Augmentation (Other): The Revision Augmentation cohort will include patients receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants during a revision surgery to correct or improve the result of a primary breast augmentation surgery.
  Interventions: Device: Mentor Siltex® Contour Profile Gel Mammary Prosthesis
- Revision Reconstruction (Other): The Revision Reconstruction cohort will include patients receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants during a revision surgery to correct or improve the result of a primary breast reconstruction surgery.
  Interventions: Device: Mentor Siltex® Contour Profile Gel Mammary Prosthesis

INTERVENTIONS:
Device: Mentor Siltex® Contour Profile Gel Mammary Prosthesis — The MENTOR® MemoryShape™ Breast Implant is a silicone elastomer mammary device with a textured surface.

SUMMARY:
The Contour Profile Gel Study is designed to demonstrate safety and effectiveness of Mentor's Mammary Prostheses in women who are undergoing primary augmentation, primary reconstruction, or revision. Safety information on the rate of capsular contracture, rupture, and infection will be collected, and used to help determine device safety.

Approximately 1000 patients at approximately 60 medical centers across the United States were enrolled in this research study. These patients were implanted with silicone breast prostheses and will be monitored for 10 years to collect information on risks associated with the implant surgery as well as changes in the way these patients feel about themselves.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring premarket approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Premarket Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A premarket approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision patients. Every patient implanted had to be part of an adjunct study, and had to be offered participation in a registry of gel-filled breast implant patients. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in a core clinical study.

In September of 2000 the Core Gel study began, leading the way to the November 2006 FDA approval of the Core Gel implant or Memory Gel breast implant.

The objective of the Contour Profile Gel Study, which started in 2002 is to determine the safety and effectiveness of the Silicone Contour Profile Gel Mammary Prostheses in women who are undergoing primary breast augmentation, primary breast reconstruction, or revision. In the duration of this study patients are required to have follow-up visits 10 weeks post-surgery and every year after surgery through the 10th year of completion. Additionally, out of the approximately 1000 patients enrolled in the CPG study, 400 have been randomly selected to have MRI scans at their 1,2,4,6,8,and 10 year post-surgery visits. Protocol changes now require all patients in this study to have MRI scans at years 6, 8, and 10.

In June of 2013 the FDA approved MENTOR® MemoryShape™ Breast Implants (CPG Style 321 Medium Height, Moderate Profile) for the following indications:

* Breast Augmentation for women at least 22 years old.
* Breast Reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subject is genetic female, 18 years of age or older
* A candidate for:

  * Primary breast augmentation (general breast enlargement)
  * Primary breast reconstruction (for trauma, loss of breast tissue due to mastectomy, malignancy, contralateral post-reconstruction symmetry, congenital deformity, including asymmetry)
  * Revision surgery (previous augmentation or reconstruction with silicone-filled or saline-filled implants)
* Signs the Informed Consent
* Agrees to return device to Mentor if explant necessary
* Agrees to comply with follow-up procedures, including returning for all follow-up visits

Exclusion Criteria:

* Subject is pregnant
* Has nursed a child within three months of study enrollment
* Been implanted with any silicone implant other than breast implants (e.g. silicone artificial joints or facial implants)
* Confirmed diagnosis of the following rheumatic diseases or syndromes: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
* Currently has a condition that could compromise or complicate wound healing (except reconstruction subjects)
* Subject in Augmentation cohort and has diagnosis of active cancer of any type. (Exception is low-grade non-metastasizing skin cancer)
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Are HIV positive
* Work for Mentor or the study doctor or are directly-related to anyone that works for Mentor or the study doctor
* Implanted metal or metal devices, history of claustrophobia or other condition that would make a MRI scan prohibitive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2002-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P Adams Jr, M.D., Principal Investigator — Dallas, TX; Dennis Hammond, M.D., Principal Investigator — Grand Rapids, MI; John Canady, M.D., Study Director — Mentor Worldwide, LLC
Locations (1):
- Mentor Worldwide, LLC, Santa Barbara, California, United States

REFERENCES:
- [Derived] Caplin DA. Indications for the use of MemoryShape breast implants in aesthetic and reconstructive breast surgery: long-term clinical outcomes of shaped versus round silicone breast implants. Plast Reconstr Surg. 2014 Sep;134(3 Suppl):27S-37S. doi: 10.1097/PRS.0000000000000609. PMID 25158767

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Augmentation: The Primary Augmentation cohort will include patients who wish general breast enlargement receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants.
  Mentor Siltex® Contour Profile Gel Mammary Prosthesis: The MENTOR® MemoryShape™ Breast Implant mammary prosthesis is a silicone elastomer mammary device with a textured surface. The Siltex® (textured) shell consists of a smooth shell bonded to an additional layer of silicone that has a textured pattern imprinted into its surface.
- Primary Reconstruction: The Primary Reconstruction cohort will include patients with loss of breast due to mastectomy or with deformities secondary to disease, malignancy, trauma, and congenital deformity receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants .
  Mentor Siltex® Contour Profile Gel Mammary Prosthesis: The MENTOR® MemoryShape™ Breast Implant mammary prosthesis is a silicone elastomer mammary device with a textured surface. The Siltex® (textured) shell consists of a smooth shell bonded to an additional layer of silicone that has a textured pattern imprinted into its surface.
- Revision Augmentation: The Revision Augmentation cohort will include patients receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants during a revision surgery to correct or improve the result of a primary breast augmentation surgery.
  Mentor Siltex® Contour Profile Gel Mammary Prosthesis: The MENTOR® MemoryShape™ Breast Implant mammary prosthesis is a silicone elastomer mammary device with a textured surface. The Siltex® (textured) shell consists of a smooth shell bonded to an additional layer of silicone that has a textured pattern imprinted into its surface.
- Revision Reconstruction: The Revision Reconstruction cohort will include patients receiving MENTOR® MemoryShape™ (formerly known as Contour Profile Gel [CPG]) Breast Implants during a revision surgery to correct or improve the result of a primary breast reconstruction surgery.
  Mentor Siltex® Contour Profile Gel Mammary Prosthesis: The MENTOR® MemoryShape™ Breast Implant mammary prosthesis is a silicone elastomer mammary device with a textured surface. The Siltex® (textured) shell consists of a smooth shell bonded to an additional layer of silicone that has a textured pattern imprinted into its surface.
Period: Overall Study
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Started | 572 | 190 | 124 | 69
Completed | 327 | 101 | 67 | 34
Not Completed | 245 | 89 | 57 | 35
Not completed — Death | 3 | 10 | 3 | 3
Not completed — Withdrawal by Subject | 14 | 12 | 8 | 2
Not completed — Lost to Follow-up | 90 | 14 | 17 | 5
Not completed — Explantation of study device(s) | 27 | 29 | 14 | 20
Not completed — Unknown reasons and patient/doctor moves | 111 | 24 | 15 | 5

BASELINE CHARACTERISTICS:
Population: All enrolled subjects are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction | Total
Number analyzed (Participants) | 572 | 190 | 124 | 69 | 955
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.58) | 47.6 (10.37) | 45.4 (9.50) | 53.2 (9.57) | 40.7 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 572 | 190 | 124 | 69 | 955
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 1 | 2 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 9 | 0 | 1 | 16
  White | 518 | 178 | 119 | 66 | 881
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 35 | 2 | 3 | 2 | 42
Region of Enrollment [Number; unit: participants]
  United States | 572 | 190 | 124 | 69 | 955

OUTCOME MEASURES:

1. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Any Reoperation
Description: Time of occurrence calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest.
Time Frame: 10 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Number analyzed (Participants) | 572 | 190 | 124 | 69
percentage of subjects | 22.3 [19.0 to 26.0] | 52.7 [45.5 to 60.2] | 35.0 [27.0 to 44.7] | 59.7 [48.0 to 71.8]

2. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Baker III, IV Capsular Contracture
Description: Baker III was identified as "firm with visible distortion" and Baker IV was identified as "obvious spherical distortion". Time of occurrence calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest.
Time Frame: 10 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Number analyzed (Participants) | 572 | 190 | 124 | 69
percentage of subjects | 3.6 [2.3 to 5.7] | 14.3 [9.6 to 21.1] | 15.5 [9.8 to 24.1] | 16.4 [9.1 to 28.5]

3. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Infection
Description: as for outcome 1
Time Frame: 10 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Number analyzed (Participants) | 572 | 190 | 124 | 69
percentage of subjects | 0.7 [0.3 to 1.9] | 1.6 [0.5 to 5.0] | 1.9 [0.5 to 7.4] | 2.9 [0.7 to 11.3]

4. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Explantation With or Without Replacement
Description: as for outcome 1
Time Frame: 10 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Number analyzed (Participants) | 572 | 190 | 124 | 69
percentage of subjects | 9.2 [7.0 to 12.0] | 34.1 [27.6 to 41.7] | 25.9 [18.7 to 35.2] | 49.0 [37.6 to 61.8]

5. Primary Outcome: Overall Mean Change in Circumferential Chest Size
Description: Change in Chest Size was calculated by subtracting the chest circumference prior to surgery from the chest circumference measured at the end of the study
Time Frame: Change from baseline to 10 years post-baseline
Population: All enrolled subjects are included.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Number analyzed (Participants) | 572 | 190 | 124 | 69
inches | 2.1 (1.69) | 0.3 (2.03) | 0.6 (1.85) | 0.1 (1.33)

ADVERSE EVENTS:
Time Frame: Baseline (Surgery) to 10 Years
Description: Adverse events were collected as Complications in alignment with 2006 FDA Guidance. Consistent with this document, complications are not classified as serious or non-serious. Key safety endpoints are summarized under Outcome Measures. All complications above 5% are reported.
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Serious Adverse Events (participants affected / at risk) | 3/572 | 10/190 | 3/124 | 3/69
Other Adverse Events (participants affected / at risk) | 91/572 | 56/190 | 20/124 | 37/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Augmentation (N=572) | Primary Reconstruction (N=190) | Revision Augmentation (N=124) | Revision Reconstruction (N=69)
Death (General disorders) | 3 | 10 | 3 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Augmentation (N=572) | Primary Reconstruction (N=190) | Revision Augmentation (N=124) | Revision Reconstruction (N=69)
Asymmetry (Surgical and medical procedures) | 4 | 19 | 4 | 3 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Baker III Capsular Contracture (Skin and subcutaneous tissue disorders) | 18 | 19 | 10 | 11 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Baker IV Capsular Contracture (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 5 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Breast Sensation Changes (Skin and subcutaneous tissue disorders) | 21 | 2 | 0 | 4 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Nipple Sensation Changes (Skin and subcutaneous tissue disorders) | 30 | 5 | 0 | 6 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Palpability-Implant (Surgical and medical procedures) | 6 | 2 | 2 | 5 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Patient Dissatisfied With Aesthetic Appearance Of Breast (Surgical and medical procedures) | 7 | 0 | 4 | 5 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Position Dissatisfaction (Skin and subcutaneous tissue disorders) | 12 | 4 | 5 | 5 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Ptosis (Skin and subcutaneous tissue disorders) | 26 | 4 | 2 | 10 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Recurrent Breast Cancer (Skin and subcutaneous tissue disorders) | 0 | 10 | 0 | 0 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.
Wrinkling (Skin and subcutaneous tissue disorders) | 15 | 9 | 8 | 8 — Complications are collected systematically using a pre-specified list of anticipated complications. Data collection did not include specification regarding each event as serious or non-serious, therefore all events are included as non-serious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and his/her collaborators are free to publish the background, methods, and results of their own research without restraint. Prior review of any proposed manuscript or abstract will be provided to the sponsor to prevent premature disclosure of trade secrets or proprietary information. The review will occur 30 days prior to submission of manuscript or abstract for consideration of publication or to a conference. Sponsor reserves right to publish or present the overall study results.